CLINICAL TRIAL: NCT06300021
Title: A Randomized, Cross-over Clinical Trial to Study the Bioavailability of Curcuminoids From Turmipure Gold® in Different Food Matrices
Brief Title: Bioavailability of Curcuminoids From Turmipure Gold® in Different Food Matrices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Givaudan France Naturals (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PEC19242; 2021-A00317-34 (Other: ID-RCB)
Record Dates: First submitted 2024-02-06; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Turmeric; Curcuminoids; Curcumin; Bioavailability; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized, cross-over, open-label, pharmacokinetic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence capsule - ready to drink - sport bar - dairy analog - gummies - probiotic drink (Experimental): Subjects receive Turmipure Gold® preparations in different food matrices in the following order: capsule - ready to drink - sport bar - dairy analog - gummies - probiotic drink
  Interventions: Dietary Supplement: TPG capsule; Dietary Supplement: TPG ready to drink; Dietary Supplement: TPG dairy analog; Dietary Supplement: TPG probiotic drink; Dietary Supplement: TPG gummies; Dietary Supplement: TPG sport bar
- Sequence dairy analog - probiotic drink - ready to drink - gummies - capsule - sport bar (Experimental): Subjects receive Turmipure Gold® preparations in different food matrices in the following order: dairy analog - probiotic drink - ready to drink - gummies - capsule - sport bar
  Interventions: Dietary Supplement: TPG capsule; Dietary Supplement: TPG ready to drink; Dietary Supplement: TPG dairy analog; Dietary Supplement: TPG probiotic drink; Dietary Supplement: TPG gummies; Dietary Supplement: TPG sport bar
- Sequence gummies - sport bar - probiotic drink - capsule - dairy analog - ready to drink (Experimental): Subjects receive Turmipure Gold® preparations in different food matrices in the following order: gummies - sport bar - probiotic drink - capsule - dairy analog - ready to drink
  Interventions: Dietary Supplement: TPG capsule; Dietary Supplement: TPG ready to drink; Dietary Supplement: TPG dairy analog; Dietary Supplement: TPG probiotic drink; Dietary Supplement: TPG gummies; Dietary Supplement: TPG sport bar
- Sequence probiotic drink - gummies - dairy analog - sport bar - ready to drink - capsule (Experimental): Subjects receive Turmipure Gold® preparations in different food matrices in the following order: probiotic drink - gummies - dairy analog - sport bar - ready to drink - capsule
  Interventions: Dietary Supplement: TPG capsule; Dietary Supplement: TPG ready to drink; Dietary Supplement: TPG dairy analog; Dietary Supplement: TPG probiotic drink; Dietary Supplement: TPG gummies; Dietary Supplement: TPG sport bar
- Sequence ready to drink - dairy analog - capsule - probiotic drink - sport bar - gummies (Experimental): Subjects receive Turmipure Gold® preparations in different food matrices in the following order: ready to drink - dairy analog - capsule - probiotic drink - sport bar - gummies
  Interventions: Dietary Supplement: TPG capsule; Dietary Supplement: TPG ready to drink; Dietary Supplement: TPG dairy analog; Dietary Supplement: TPG probiotic drink; Dietary Supplement: TPG gummies; Dietary Supplement: TPG sport bar
- Sequence sport bar - capsule - gummies - ready to drink - probiotic drink - dairy analog (Experimental): Subjects receive Turmipure Gold® preparations in different food matrices in the following order: sport bar - capsule - gummies - ready to drink - probiotic drink - dairy analog
  Interventions: Dietary Supplement: TPG capsule; Dietary Supplement: TPG ready to drink; Dietary Supplement: TPG dairy analog; Dietary Supplement: TPG probiotic drink; Dietary Supplement: TPG gummies; Dietary Supplement: TPG sport bar

INTERVENTIONS:
Dietary Supplement: TPG capsule — A dietary supplement product in capsule form containing 300 mg Turmipure Gold®
Dietary Supplement: TPG ready to drink — Ingredient stick containing 300 mg Turmipure Gold® mixed in 60 mL mango fruit nectar
Dietary Supplement: TPG dairy analog — Ingredient stick containing 300 mg Turmipure Gold® mixed in 240 mL oat milk
Dietary Supplement: TPG probiotic drink — Ingredient stick containing 300 mg Turmipure Gold® mixed in a 100 mL probiotic yogurt drink base
Dietary Supplement: TPG gummies — Pectin gummies containing 300 mg Turmipure Gold®
Dietary Supplement: TPG sport bar — Sport nutrition bar containing 300 mg Turmipure Gold®

SUMMARY:
The goal of this clinical trial is to learn about the extent to which turmeric compounds in different food matrices becomes available to the body in healthy volunteers. The main question it aims to answer is:

* Is the availability to the body of a turmeric dietary supplement altered when consumed in fruit nectar, oat milk, yogurt drink, or gummies in comparison to a dietary supplement capsule?

Participants will ingest a turmeric dietary supplement as a capsule or in different food matrices on six testing days (separated by at least one week). The day before testing day, a standardized dinner will be provided to the participants in the evening and participants will be instructed to not consume any foods or beverages (except water) and to arrive fasted (12 hours) at the investigation site. Participants will ingest turmeric dietary supplement formulations one by one in random order in the morning of testing days. Regular blood and urine samples will be collected before and up to 24 hours after the turmeric dietary supplement ingestion. Standardized meals will be provided during the entire testing day (lunch, mid-afternoon snack, dinner).

DETAILED DESCRIPTION:
Curcumin has been studied as the main bioactive component of the rhizome of the herb Curcuma longa, known as turmeric, and is associated to potential health effects and benefits. Other bioactive components have also been identified, called the curcuminoid group. Curcuminoids are natural yellow-orange pigments and hydrophobic polyphenols derived from. Extracts of turmeric generally contain 75-80% curcumin, 15-20% demethoxycurcumin (DMC), and 0-10% bisdemethoxycurcumin (BDMC). Curcumin and curcuminoids have been extensively investigated due to their antioxidant and anti-inflammatory properties, notably regarding their potential efficacy in modulating various health conditions.

In the present trial, the aim is to assess the bioavailability of curcuminoids in different food matrix formulations, the capsule format being the reference matrix, with a hypothesis of equivalence. The primary objective of the study is to assess the plasmatic concentration profile of total curcuminoids (curcumin, DMC, BDMC and their metabolites) on a 24-hour period after consumption of five different food matrix formulations containing TPG in comparison to the dietary supplement capsule formulation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years (limits included)
* BMI between 18.5 and 24.9 kg/m² (limits included)
* Weight stable within ±3 kg in the last three months
* With routine blood chemistry values within the normal range
* For women: Non menopausal with the same reliable contraception since at least 3 cycles before the beginning of the study and agreeing to keep it during the entire duration of the study or menopausal without or with hormone replacement therapy since at least 3 months
* Non-smoking or with tobacco consumption ≤5 cigarettes per day and agreeing not to smoke during the entire duration of the study
* Good general and mental health in the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by dated and signed informed consent form
* Affiliated with a social security scheme
* Agreeing to be registered on the volunteers in biomedical research file

Exclusion Criteria:

* Suffering from a metabolic or endocrine disorder such as diabetes, uncontrolled or controlled thyroidal trouble or other metabolic disorder
* Suffering from a chronic disease (e.g. cancer, HIV, kidney failure, ongoing hepatic or biliary disorders, chronic inflammatory digestive disease, arthritis, anemia or other chronic respiratory trouble, gammapathies, hepatic diseases, decompensated diabetes, tuberculosis, ulcerative colitis, parkinson's disease, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease)
* Suffering from liver diseases
* Having medical history of current pathology which could affect the study results or expose the subject to an additional risk according to the investigator (IBS, chronic diarrhea, constipation or abdominal pain, inflammatory bowel diseases (Crohn's disease or ulcerative colitis), cirrhosis, chronic laxatives use, severe COVID-19 history (requiring oxygen-therapy) in the 12 past months, …)
* Recent gastroenteritis or food borne illness such as confirmed food poisoning (less than 1 month)
* With a low venous capital of blood samples according to the investigator's opinion
* With a known or suspected allergy or intolerance to any food
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient or turmeric and/or of the standard meals
* Pregnant or lactating women or intending to become pregnant within 3 months ahead
* Currently taking any chronic drug treatment (for example: antidiabetics, anticoagulant, antihypertensive treatment, treatment thyroid, asthma treatment, anxiolytic, antidepressant, lipid-lowering treatment, corticosteroids, phlebotonic, veinotonic, drug with impact on blood circulation, …) except oral and local contraceptives,
* Currently taking or having taken any supplementation from botanical origins or with curcumin in the previous 3 months before inclusion
* Currently taking or having taken laxatives or antibiotics, in the previous 3 months before the V0 visit
* Currently taking or having taken any prebiotics or probiotics supplementation from food or from dietary supplements in the previous 3 months before the V0 visit
* With significant change in food habits or in physical activity in the 3 months before the V0 visit or not agreeing to keep them unchanged throughout the study
* Trying to lose weight with a current or planned in the next 3 months specific diet (hyper- or hypocaloric, vegan, vegetarian, …) or exercise regimen
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator
* Exhibiting alcohol or consuming more than 3 standard drinks of alcoholic beverage daily for men or 2 daily for women or not agreeing to keep alcohol consumption habits unchanged throughout the study or drug dependence or exhibiting drug dependence
* Having a lifestyle deemed incompatible with the study according to the investigator including high level physical activity (defined as more than 5 hours of significant physical activity a week, walking excluded)
* Having taken part in another clinical trial in the previous 3 months or being in the exclusion period of a previous clinical trial
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros
* Under legal protection (guardianship, wardship) or deprived from rights following administrative or judicial decision
* Presenting a psychological or linguistic incapability to sign the informed consent
* Impossible to contact in case of emergency
* Having consumed curcumin-containing food supplements (curcumin, turmeric and curry) or foods (curcumin, turmeric, E100, and curry) defined as at least 3 times per week and for 2 weeks prior to testing
* Made a blood donation in the 3 months before the V0 visit or intending to make it within 3 months ahead
* After V0 biological analyses the subject will be considered as non-eligible to the study on the following criteria: Control record (glycaemia, total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol, GGT, ASAT, ALAT, urea, creatinine, total bilirubin and CBC) with clinically significant abnormality according to the investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Dose-normalized AUC0-24h of total curcuminoids | 0 to 24 hours
  Normalized (according to mg of curcuminoids ingested) area under the concentration-time curve from 0 to 24 h of total curcuminoids (sum of all quantified metabolites) in plasma:
  * Total curcuminoids = curcumin + demethoxycurcumin (DMC) + bisdemethoxycurcumin (BDMC) + tetrahydrocurcumin (THC) + hexahydrocurcumin (HHC) + curcumin glucuronide + DMC glucuronide + BDMC glucuronide + THC glucuronide + HHC glucuronide + curcumin sulfate + DMC sulfate + BDMC sulfate + THC sulfate + HHC sulfate

SECONDARY OUTCOMES:
Dose-normalized AUC0-24h of curcuminoid compounds and of their metabolites | 0 to 24 hours
  Normalized (according to mg of curcuminoids ingested) area under the plasma concentration-time curve from 0 to 24 h of:
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites
Dose-normalized AUC0-8h of total curcuminoids, curcuminoid compounds and of their metabolites | 0 to 8 hours
  Normalized (according to mg of curcuminoids ingested) area under the plasma concentration-time curve from 0 to 8 h of:
  * Total curcuminoids
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites
Dose-normalized AUC0-∞ of total curcuminoids, curcuminoid compounds and of their metabolites | Data collected from 0 to 24 hours
  Normalized (according to mg of curcuminoids ingested) area under the plasma concentration-time curve from 0 hours to extrapolated infinite time of:
  * Total curcuminoids
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites
AUC0-24h of total curcuminoids, curcuminoid compounds and of their metabolites | 0 to 24 hours
  Area under the plasma concentration-time curve from 0 to 24 h of:
  * Total curcuminoids
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites
AUC0-8h of total curcuminoids, curcuminoid compounds and of their metabolites | 0 to 8 hours
  Area under the plasma concentration-time curve from 0 to 8 h of:
  * Total curcuminoids
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites
AUC0-∞ of total curcuminoids, curcuminoid compounds and of their metabolites | Data collected from 0 to 24 hours
  Area under the plasma concentration-time curve from 0 hours to extrapolated infinite time of:
  * Total curcuminoids
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites
Relative bioavailability for normalized AUC0-24h of total curcuminoids, curcuminoid compounds and of their metabolites | 0 to 24 hours
  Relative bioavailability (ratio of the dose-normalized AUCs) in different food matrices versus capsule format of:
  * Total curcuminoids
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites
Relative bioavailability for normalized AUC0-8h of total curcuminoids, curcuminoid compounds and of their metabolites | 0 to 8 hours
  Relative bioavailability (ratio of the dose-normalized AUCs) in different food matrices versus capsule format of:
  * Total curcuminoids
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites
Relative bioavailability for normalized AUC0-∞ of total curcuminoids, curcuminoid compounds and of their metabolites | Data collected from 0 to 24 hours
  Relative bioavailability (ratio of the dose-normalized AUCs) in different food matrices versus capsule format of:
  * Total curcuminoids
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites
Cmax of total curcuminoids, curcuminoid compounds and of their metabolites | 0 to 24 hours
  Peak plasma concentration of:
  * Total curcuminoids
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites
Dose-normalized Cmax of total curcuminoids, curcuminoid compounds and of their metabolites | 0 to 24 hours
  Normalized (according curcuminoids ingested) peak plasma concentration of:
  * Total curcuminoids
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites
Half-life of total curcuminoids, curcuminoid compounds and of their metabolites | 0 to 24 hours
  Time after which the plasma concentration decreased by half of:
  * Total curcuminoids
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites
Tmax of total curcuminoids, curcuminoid compounds and of their metabolites | 0 to 24 hours
  Time to peak plasma concentration of:
  * Total curcuminoids
  * Total parent compounds
  * Total sulfate metabolites
  * Total glucuronide metabolites
  * Total parent compounds and their relative sulfate and glucuronide metabolites
  * Curcumin and its relative sulfate and glucuronide metabolites
  * DMC and its relative sulfate and glucuronide metabolites
  * BDMC and its relative sulfate and glucuronide metabolites
  * Curcumin and all its relative metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Metreau, MD, Principal Investigator — BioFortis
Locations (1):
- Biofortis, Saint-Herblain, France